CLINICAL TRIAL: NCT05245422
Title: Parent And Infant Relief (PAIR): Acceptance of a Partially Hydrolyzed Formula
Brief Title: Acceptance of a Partially Hydrolyzed Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3392-1
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Fussy Infant (Baby)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cow's milk intact protein infant formula (Active Comparator): Control
  Interventions: Other: Infant Formula - Intact protein
- Partially hydrolyzed cow's milk protein infant formula (Experimental): Investigational
  Interventions: Other: Infant Formula - Partially hydrolyzed protein

INTERVENTIONS:
Other: Infant Formula - Partially hydrolyzed protein — Partially hydrolyzed cow's milk protein
  Arms: Partially hydrolyzed cow's milk protein infant formula
Other: Infant Formula - Intact protein — Intact cow's milk protein
  Arms: Cow's milk intact protein infant formula

SUMMARY:
A multi-center, double-blind, controlled, parallel-designed, prospective trial intended to evaluate the nutritive effects of a partially hydrolyzed cow's milk protein infant formula on infant fussiness.

DETAILED DESCRIPTION:
A multi-center, double-blind, controlled, parallel-designed, prospective trial intended to evaluate the nutritive effects of a partially hydrolyzed cow's milk protein (PHP) infant formula on infant fussiness. Formula tolerance and intake, sleep characteristics, stool characteristics, parental quality of life, and medically confirmed adverse events will be compared between i two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver has reliable access to the internet and a reliable device (such as a computer, tablet, or smartphone) to access mobile apps and be able to view and complete study questionnaires
* Singleton birth
* 15 to 75 days of age at Visit 1, inclusive (day of birth is considered Day 0)
* Gestational age of ≥37 to 42 weeks (36 weeks and six days is considered 36 weeks' gestational age)
* Birth weight of 2500 g (5 lbs 8 oz) or more
* Exclusively receiving an intact protein infant formula (cow's milk-based or plant-based) for 7 days prior to Visit 1
* Answer to question: "On average, how fussy has your baby been over the past 3 days" is moderately fussy, very fussy, or extremely fussy at Visit 1
* Parent(s) or legal guardian has full intention to exclusively feed study formula during the study period
* Parent(s) or legal guardian agrees not to enroll infant in another interventional clinical study while participating in this study
* Signed informed consent obtained from parent or legal guardian for infant's participation in the study
* Signed authorization obtained from parent or legal guardian to use and/or disclose Protected Health Information for infant from birth through the length of the study period

Exclusion Criteria:

* Infant has been weighed by a health care professional (HCP) and is identified with inadequate weight gain or failure-to-thrive
* Diagnosis or suspicion of cow's milk protein allergy by a healthcare professional
* Any acute illness within the 3 days prior to Visit 1
* Infant has had immunizations or a surgical procedure within the 3 days prior to or on Visit 1
* Immunizations are planned for the infant during any of the 7 days after Visit 1
* Use of oral, intramuscular or intravenous antibiotics within the 7 days prior to Visit 1
* Infant has had bloody stools (visible to the naked eye) within the 7 days prior to Visit 1
* Infant has been taking medication (prescribed and over-the-counter) for gastrointestinal conditions for any of the 7 days prior to Visit 1 (however, probiotics are allowed)
* Infant has a surgical procedure planned during the study period
* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* History of underlying neurological or organic disease likely to cause fussiness, such as (but not limited to) a doctor's diagnosis of neonatal abstinence syndrome and inflammatory or orthopedic disorders
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as combined immunodeficiencies, DiGeorge syndrome, Wiskott-Aldrich syndrome, severe congenital neutropenia and secondary immunodeficiencies linked to HIV infection, Down syndrome or others)

Ages: 15 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Fussiness | Study Feeding Days 1 through 7
  Daily Diary

SECONDARY OUTCOMES:
Fussiness | Study Feeding Days 8-28
  Daily Diary
Gassiness | Study Feeding Days 1-28
  Daily Diary
Crying | Study Feeding Days 1-28
  Daily Diary
Spit-up | Study Feeding Days 1-28
  Daily Diary
Sleep | Study Feeding Days 1-28
  Daily Diary
Stool frequency | Study Feeding Days 1-28
  Daily Diary
Stool consistency | Study Feeding Days 1-28
  Daily Diary
Study Formula Intake | Study Feeding Day 7 and Study Feeding Day 25 (+3 days)
  24-hour Recall of Study Formula Intake
Brief Infant Sleep Questionnaire | Study Feeding Day 14 (+2 days) and Study Feeding Day 25 (+ 3 days)
  Revised Short Form (BISQ-R SF)
Quality of Life Questionnaire | Study Feeding Day 7 (+2 days) and Study Feeding Day 25 (+3 days)
  Pediatric Quality of Life Inventory™ Family Impact Module (PedsQL FIM)-Acute
Medically confirmed adverse events | Day 1 through end of feeding
  Collected from medical records

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - DBC Research USA, Miramar, Florida
  - Proactive Clinical Research, Sarasota, Florida
  - Mid Valley Research Inc., Moline, Illinois
  - Frontier Pediatric Research, Lincoln, Nebraska
  - Meridian Clinical Research, Charleston, South Carolina
  - Tribe Clinical Research, Greenville, South Carolina
  - AVIATI Healthcare & Clinical Research, Memphis, Tennessee
  - South Texas Pediatric Research Group, Del Rio, Texas
  - Proactive Clinical Research, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabrizio V, Bohan Brown MM, Boucher P, Boyd S, Cao S, Davis C, Johnson S, Khan N, Moore N, Muse K, Ogwara F, Patterson AC, Wampler JL, Yeiser M, Zhuang W, Wu SS. A Randomized Controlled Trial of a Partially Hydrolyzed Formula on Comfort Measures in Fussy Infants. Curr Dev Nutr. 2025 Oct 13;9(11):107574. doi: 10.1016/j.cdnut.2025.107574. eCollection 2025 Nov. PMID 41323693